CLINICAL TRIAL: NCT01292551
Title: Treatment With Endothelin Antagonist to Tcpc Patients; a Multicenter, Randomized, Prospective Study Measuring Maximal O2 Uptake in Ergometer Bicycle Test
Brief Title: Study of Placebo or Bosentan to Treat Patients With Single Ventricle Physiology.
Acronym: TEMPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Bispebjerg Hospital (Other); Actelion (Industry)
Responsible Party: Principal Investigator, Anders Hebert, M.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEMPO study; 2010-022389-28 (EudraCT Number)
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Hypoplastic Left Heart Syndrome; Tricuspid Atresia; Other Specified Congenital Anomalies of Heart
Keywords: single ventricle physiology; Fontan procedure
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Tricuspid Atresia | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bosentan (Active Comparator)
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — tablets Bosentan 62,5 mg x 2 daily for two weeks, then 125 mg x 2 daily for 12 weeks
  Other Names: Bosentan: Tracleer
  Arms: Bosentan
Drug: Placebo — Placebo tablets 2 x daily for 2 weeks, then change to different placebo tablets to match Bosentan group, 2 x daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Bosentan is an effective and safe treatment to adolescent and adult (15 years and older) patients, born with one ventricle of the heart instead of two (single ventricle physiology) and who have undergone TCPC as a palliative surgical treatment. The aim of the TCPC operation is to use the one functioning ventricle to pump the blood flow to the body, while the blood to the lungs is received directly from the caval veins, and is thus a passive flow, without the aid of a ventricle to actively pump the blood through the pulmonary circulation. The resistance in the pulmonary circulation is therefore critical to these patients. These patients have markedly lower work capacity in bicycle test than the general public. Furthermore they have a high risk of developing complications e.g. loss of protein from the intestines.

Bosentan is a medication that lowers the resistance in the pulmonary circulation. It is routinely used for patients with pulmonary hypertension. Some studies have shown that drugs that lower the pulmonary resistance can increase exercise capacity significantly in patients with single ventricle physiology.

In this study 80 patients will receive either placebo or Bosentan for 14 weeks. Before and after the treatment, bicycle test along with blood samples, stool samples and quality of life interviews will be performed. Every four weeks during the study blood samples, physical exam and interviews will be performed to ensure the safety of the treatment.

The investigators expect to find a significant increase in work capacity after 14 weeks in the treatment group compared with the placebo group.

Moreover the investigators hope to find a decrease in intestinal protein loss and an improved quality of life.

DETAILED DESCRIPTION:
In the statistical analysis the investigators wish to analyse interactions between the primary endpoint and predefined subgroups in order to distinguish responders from non-responders to the treatment. The predefined subgroups are:

NT-proBNP > 100 (yes/no) Ventricular anatomy (RV/LV) CT-proEndothelin-1. In the latter, the investigators do not wish to predefine a specific value, due to limited experience with this analysis. We wish to use the data from the study to find a cut-off value, that is able to predict positive response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* TCPC operated
* Age > 15 years old
* Clinical stability > 3 months, evaluated by investigator from clinical record
* For women: Negative s-hCG and use of contraception

Exclusion Criteria:

* Severe heart failure (NYHA-class IV)
* Oxygen saturation < 85 % at rest
* Pre-existing liver condition (transaminases 2x > reference)
* Renal failure (creatinin > 150 mmol/l)
* Obstruction of TCPC circulation
* History of work induced severe arrhythmia
* Systolic blood pressure below 80% of reference (BT < 88 mmHg)
* Use of any of following drugs: Fluconazol, Ketoconazole, CiclosporinA, Lopinavir, Ritonavir, Rifampicin, Carbamazepin and Phenytoin
* Significant extra-cardiac condition e.g. neurological impairment

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in VO2max at 14 weeks | Baseline and 14 weeks
  Maximal O2 uptake in ml/min/kg in ergometer bicycle test

SECONDARY OUTCOMES:
Change from baseline in blood samples at 14 weeks | Baseline and 14 weeks
  blood samples measured: plasma CT pro endothelin-1, IgG, IgA, NT pro BNP, albumin, free protein
Change from baseline in SF36 questionnaire score at 14 weeks | Baseline and 14 weeks
  SF36 quality of life interview
Change from baseline in feces alfa 1 antitrypsin at 14 weeks | Baseline and 14 weeks
  Fecal alfa 1 antitrypsin in mg/g
Number of participants with adverse events | 2, 6, 10 and 14 weeks after start of treatment
  general interview on adverse effects, and questions with special focus on typical adverse effects in Bosentan
Change from baseline in vital signs | Baseline, 2, 6, 10 and 14 weeks
  Systemic bloodpressure in mmHg, Pulse in min-1, Oxygen saturation in percent
Change from baseline in control blood samples | Baseline, 2, 6, 10 and 14 weeks
  Liver and renal biomarkers, Hb, PCV, trc and hCG for women
Change from baseline in cardiac output/pulmonary blood flow | Baseline and 14 weeks
  CO measured by Stringer Wassermann method during ergometer bicycle test

CONTACTS AND LOCATIONS:
Overall Officials: Lars Sondergaard, DMSc, Study Director — Rigshospitalet, Denmark; Anders H Hebert, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (4):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska Institutet, Stockholm

REFERENCES:
- [Derived] Hebert A, Mikkelsen UR, Thilen U, Idorn L, Jensen AS, Nagy E, Hanseus K, Sorensen KE, Sondergaard L. Bosentan improves exercise capacity in adolescents and adults after Fontan operation: the TEMPO (Treatment With Endothelin Receptor Antagonist in Fontan Patients, a Randomized, Placebo-Controlled, Double-Blind Study Measuring Peak Oxygen Consumption) study. Circulation. 2014 Dec 2;130(23):2021-30. doi: 10.1161/CIRCULATIONAHA.113.008441. Epub 2014 Oct 20. PMID 25446057
- [Derived] Hebert A, Jensen AS, Idorn L, Sorensen KE, Sondergaard L. The effect of bosentan on exercise capacity in Fontan patients; rationale and design for the TEMPO study. BMC Cardiovasc Disord. 2013 May 11;13:36. doi: 10.1186/1471-2261-13-36. PMID 23663658